CLINICAL TRIAL: NCT06133738
Title: The Effectiveness of an Internet-Based Cognitive Behavioural Therapy and Exercise in Chronic Knee Patients With Psychological Distress: Clinical Trail Protocol
Brief Title: Effects of iCBT and Exercise for Chronic Knee Patients
Acronym: iCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bahrain (Other)
Responsible Party: Principal Investigator, Amal Alaradi, Senior Physiotherapist, University of Bahrain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iCBTExCKP
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Chronic Knee Pain
Keywords: Internet Based Cognitive Behavioural Therapy; Psychological Distress; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This will be a 2-arm quasi-randomized controlled trial of eight weeks of intervention involving eight sessions of standardized exercise program and either concomitant iCBT and educational sessions or educational sessions only. Measurements will be taken at baseline and eight weeks immediately following the intervention. Primary outcome measures are a numerical pain rating scale, 40-m Fast-Paced Walk Test, Step Test, and 30 seconds Chair Stand Test. Secondary outcome measures are Patient Health Questionnaire, Psychological Distress, Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form, Health-Related Quality of Life-Short Form-12, and Quadriceps Maximum Isometric Muscle Strength.
Who Masked: Participant
Masking Description: Eligible patients will be randomly allocated to either the study group or the control group (1:1). Participants will be blinded to their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will be given 8 sessions of a standardized exercise program, a link to access online educational sessions, in addition to internet based cognitive behavioural therapy sessions.
  Interventions: Other: Standardized Exercise Program; Other: Internet based Cognitive Behavioral Therapy; Other: Educational Materials
- Control Group (Active Comparator): Participants in this group will be given 8 sessions of a standardized exercise program and a link to access online educational sessions.
  Interventions: Other: Standardized Exercise Program; Other: Educational Materials

INTERVENTIONS:
Other: Standardized Exercise Program — Participants will be asked to attend to the department for 8 supervised physiotherapy sessions designed to strengthen lower limb muscles. Eight sessions were chosen as this number should be able to achieve improvements in pain and function. Standardized exercises sessions will be held once weekly in the health center and will be supervised by the researcher. In addition, participants will be requested to perform the prescribed exercises 3 times per week at home, with 1-2 days rest interval between the exercise's sessions.
  The program is comprised of a minimum of 4 and a maximum of 6 individualized lower limb exercises to be performed 4 times per week (once in the health center and 3 times at home). All exercise programs will include at least 2 knee extensor strengthening exercises, 1 hip abductor strengthening exercise, 1 hamstring strengthening exercise, 1 calf strengthening exercise, and 1 other exercise will be chosen based on assessment findings.
Other: Internet based Cognitive Behavioral Therapy — This intervention will be given to participants in intervention group. This is a link to access pre-recorded online sessions of CBT.
  The iCBT link contained eight 35- to 45-minute sessions, designed to be completed weekly, each provided an explanation of a cognitive or behavioural pain coping skill. Session 1 provided an overview, including a therapeutic rationale of CBT, followed by training in progressive muscle relaxation. Sessions 2 through 7 taught brief relaxation skills, activity-rest cycling, pleasant activity scheduling, cognitive restructuring, pleasant imagery, and problem-solving. Session 8 consolidated the learnt and taught strategies for long-term skill use. Each session has to be completed within the same week where the physiotherapy session is given.
  The researcher has developed a website that contained all the CBT materials.
  Arms: Intervention Group
Other: Educational Materials — All participants will receive a link to access online educational material about chronic knee pain. This is a YouTube link that consists of 5 sessions, with each lasting for 5-7 minutes, and is comprised of general information about the following: healthy eating, osteoarthritis and X-Ray, physical activity, the full pain experience, and proper footwear. Participants will be encouraged to access the educational material at their own leisure and pace.

SUMMARY:
The goal of this clinical trial is to study the effects of using an internet-based cognitive behavioural therapy (iCBT) program and exercise in chronic knee patients with psychological distress. The main question[s] it aims to answer are:

* What are the effects of a combined iCBT and standardized exercise program on pain and function in chronic knee pain patients with psychological distress
* What are the effects of a combined iCBT and standardized exercise program on depression, psychological distress, physical function, quality of life, and quadriceps muscle strength in chronic knee pain patients with psychological distress
* Do a combined iCBT and standardized exercise program significantly improve pain and function in chronic knee pain patients with psychological distress compared to a control group?
* Do a combined iCBT and standardized exercise program significantly improve depression, psychological distress, physical function, QoL, and quadriceps muscles strength in chronic knee pain patients with psychological distress compared to a control group?

Participants will be allocated randomly to either intervention group or control group.

Intervention group will be given iCBT, exercise and educational program, while the control group will be given exercise and educational program only.

Researchers will compare both groups to see if the intervention group improves much better in terms of pain, function and other outcome measures compared to the study group.

DETAILED DESCRIPTION:
This will be a 2-arm quasi-randomized controlled trial of eight weeks of intervention involving eight sessions of standardized exercise program and either concomitant iCBT and educational sessions or educational sessions only. Measurements will be taken at baseline and eight weeks immediately following the intervention. Primary outcome measures are a numerical pain rating scale, 40-m Fast-Paced Walk Test, Step Test, and 30 seconds Chair Stand Test. Secondary outcome measures are Patient Health Questionnaire, Psychological Distress, Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form, Health-Related Quality of Life-Short Form-12, and Quadriceps Maximum Isometric Muscle Strength.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years
2. Depression level of at least 2 out 6 on the PHQ-2 questionnaire and/or psychological distress level (K-6) of at least 7 out of 24
3. Knee pain for more than 3 months and for most days of the previous month
4. A minimum average knee pain intensity of 4 on an 11-point numeric rating scale in the previous week
5. Mild to moderate difficulty with physical activities on KOOS-PS questionnaire, at least 6 out of 24
6. Has a smartphone with internet access.

Exclusion Criteria:

1. Knee surgery including arthroscopy within the past 6 months
2. Awaiting or planning any back or lower limb surgery within the next 12 months
3. Current or past (within 3 months) oral or intra-articular corticosteroid use
4. Current long-term use of analgesics or drugs that cause analgesic effects such as the drugs used for epilepsy and bipolar disorders
5. Systemic arthritic conditions such as rheumatoid arthritis
6. Physiotherapy, chiropractic or acupuncture treatment or exercises specifically for the knee within the past 6 months
7. Walking >30 min continuously daily or participating in a regular (more than twice a week) exercise program
8. Past participation in a CBT program
9. Inability to walk unaided as this is necessary for some of the physical testing
10. Grade IV on Kellgren and Lawrence grading system for Osteoarthritis classification
11. Medical condition precluding safe exercise such as uncontrolled hypertension or heart condition
12. Major joint pain (e.g., back, hip or ankle) to a greater extent than the knee pain that could limit the ability to exercise
13. Self-reported psychiatric history such as schizophrenia, epilepsy, and bipolar disorders
14. Self-reported diagnosis of current clinical depression
15. Neurological condition such as Parkinson's disease, Multiple sclerosis, or stroke
16. Inadequate written and spoken Arabic
17. Unable to comply with the protocol such as the inability to attend therapy sessions or attend assessment appointments at the health center.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The Single-Item Numerical Rating Scale (NRS) | 8 weeks
  Participants will be asked to rate their average knee pain in the past week on a scale from 0 to 10, with '0' meaning 'No pain' and '10' meaning 'Pain as bad as you can imagine'. This will be recorded via online form.
40-m Fast-Paced Walk Test (40-m FPWT) | 8 weeks
  A participant will be instructed to walk as quickly but as safely as possible to a mark 10 m away, return, and repeat for a total distance of 40 m. Time of one trial, with turn time excluded, will be recorded and expressed as speed m/s by dividing distance (40 m) by time (s).
Step Test (ST) | 8 weeks
  This test will be performed while the participant maintains balance on the study limb, then the contralateral foot will be stepped on and off a 15-cm step as many times as possible within 15 seconds. The count of the number of times the participant could step the foot up and return it to the floor over a 15-s interval will be recorded. The test will performed with no hand support allowed. For participants with unilateral knee OA, the test will be performed while standing on the affected side. For participants with bilateral knee OA, the most symptomatic limb will be considered the osteoarthritic limb for the purpose of this study.
30 seconds Chair Stand Test (30s CTS test) | 8 weeks
  From the sitting position in the middle of seat with feet shoulder-width apart, ﬂat on the ﬂoor, arms crossed at chest, a participant will be asked to stand completely up, then sit completely back down, repeatedly for 30s. The chair will be against a wall. Count the total number of complete chair stands (up and down represents one stand) of one trial. If a full stand is completed at 30s then this is counted in the total. The same chair is used for re-testing.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-2) | 8 weeks
  This is a 2-item scale for depression screening in primary care. This questionnaire will be administered via online forms. A PHQ-2 score ranges from 0-6, with 0 indicating the lowest level of depression, and 6 indicating the highest level of depression.
Psychological Distress (Kessler 6) | 8 weeks
  This is a 6-item self-report questionnaire that measures psychological distress based on anxiety and depressive symptoms in the patient's most recent 4-week period. The range for summed responses on the K6 Scale is 0 to 24, with 0 suggesting the lowest level of nonspecific psychological distress, and 24 suggesting the highest level of nonspecific psychological distress. This questionnaire will be administered via online forms.
Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS- PS) | 8 weeks
  This is a 7-item measure of physical function derived from the items of the Function, daily living and Function, sports, and recreational activity subscales of the KOOS. It will be administered through an online survey. The range for summed responses on the KOOS-PS is 0 to 24, where 24 is the worst possible and 0 is the best possible score. This questionnaire will be administered via online forms.
Health-Related Quality of Life-Short Form-12 (SF-12) | 8 weeks
  This is a questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health-related QoL. Scores range from 0 to 50, with higher scores indicating better health status. It will be administered through an online survey.
Maximum Isometric Muscle Strength | 8 weeks
  Maximal voluntary isometric quadriceps muscle strength will be assessed using a hand-held dynamometer. To do the test, a participant is seated on an examination table with their knees flexed to 60° and their feet off the ground. The hand-held dynamometer is positioned on the anterior aspect of the distal tibia, just superior to the malleoli. The participant grasps the examination table with his/her hands for stabilization, and the participant is instructed to extend his/her knee "as hard as possible" into the hand-held dynamometer. The participant continues to exert force into the hand-held dynamometer for 4 s, and the maximum force across the trial is recorded. Three testing trials will be completed, and the average force (Newtons [N]) across the three trials will be normalized to body mass (N/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Alaradi, Principal Investigator — Primary Healthcare Centers- Kingdom of Bahrain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT06133738/Prot_SAP_000.pdf